CLINICAL TRIAL: NCT03741868
Title: Symptom Burden and Unmet Supportive Care Needs in Lung Cancer Patients Undergoing First or Second Line Immunotherapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Lung Cancer Initiative of North Carolina (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00046256; CCCWFU01517 (Other: Wake Forest Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Lung Neoplasm
Keywords: Lung Cancer; Immunotherapy; Stage IV cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage IV non-small cell lung cancer: 60 - stage IV non-small cell lung cancer patients will be recruited through the Wake Forest Baptist Comprehensive Cancer Center to complete the quantitative portion of the study. We will use purposive sampling to assure representation of patients at different stages in immunotherapy (i.e., initiating treatment, anticipating scan results, after onset of immune-related side effects).12-15 of the 60 patients who complete the survey and who express interest in providing feedback on programs and participating in future research will be recruited to complete the qualitative portion of the study

SUMMARY:
Doctors are recruiting patients receiving care for lung cancer at the Wake Forest Baptist Comprehensive Cancer Center asking about needs and experiences during immunotherapy. Immunotherapy is a new treatment for lung cancer. The research is to better understand patients' perspectives on what immunotherapy is like and will provide important information to help understand the symptoms patients experience, the impact of treatment on daily life, ways that people adapt to the challenges of treatment, and services that may help people live better during treatment.

DETAILED DESCRIPTION:
The overall primary objective of this pilot study is to describe patient-reported symptom burden, unmet supportive care needs, and use of and interest in supportive care services in stage IV non-small cell lung cancer patients undergoing first or second line immunotherapy and to identify psychosocial factors associated with these outcomes.

60 stage IV non-small cell lung cancer patients will be recruited through the Wake Forest Baptist Comprehensive Cancer Center. The study team will use purposive sampling to assure representation of patients at different stages in immunotherapy (i.e., initiating treatment, anticipating scan results, after onset of immune-related side effects).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV (per AJCC 7th edition) non-small cell lung cancer.
* Receiving first or second line immunotherapy.
* ECOG Performance status of 0-3.
* English-speaking

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Women of all races and ethnicity who meet the above-described eligibility criteria are eligible for this trial.
  * Based on WFBCCC population estimates, we expect approximately 41% of participants to be women. Translating this to our sample size estimate of 60, we plan to enroll at least 25 women. Similarly, we expect approximately 1% of study participants to be Hispanic/Latin. 10% Black or African American, 1% American Indian/Alaska Native, 1% Asian. .
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
NCI-PRO-CTCAE items | Past 7 days prior to completion of survey
  The NCI-PRO-CTCAE questionnaire will measure patient reported immune-mediated side effect frequency, severity, and interference of selected symptoms on a varied 1-5 scale with lower scales denoting better outcomes. Higher scores reflect greater symptom severity
PROMIS Fatigue | Past 7 days prior to completion of survey
  The PROMIS Fatigue questionnaire will measure patient reported fatigue on a varied 1-5 scale with lower scales denoting better outcomes. 8 items responded to on a 1-5 likert type scale, with higher scores reflecting greater fatigue.
EORTC-QLQ-30 questionnaire | Past 7 days prior to completion of survey or 7 days after completion of survey
  EORTC-QLQ-30 questionnaire will measure the patient-reported disease and treatment related symptom severity and interference of 5 functional subscales and 9 symptom subscales. Items are rated on a four-point scale with 1 = not at all to 4 = very much. Subscales are transformed linearly to have a range of 0-100, with higher scores reflecting better function on the 5 functional scales or a higher symptom burden on the symptom scales
Functional Assessment of Chronic Illness Therapy - Comprehensive Score for Financial Toxicity (FACIT-COST) | Past 7 days prior to completion of survey
  The FACIT-COST will measure patient reported financial toxicity on a 0 (not at all) - 4 (very much) scale with higher scores denoting better outcomes. Scores calculated following the FACIT scoring procedures such that a higher score represents less financial distress.
Supportive Care Needs Survey-Short Form 34 (SCNSF34) questionnaire | Past 30 days prior to completion of survey
  The Supportive Care Needs Survey-Short Form 34 questionnaire will measure unmet supportive care needs with a scale of 1 (not applicable) to 5 (high need) with lower score indicating better outcome. Responses are provided on a divided 5-point Likert scale (no unmet need indicated by 1 = not applicable or 2 = satisfied; unmet need indicated by 3 = low need, 4 = moderate need, or 5 = high need). The measure contains 5 domains: health system and information, patient care and support, physical and daily living, psychological, and sexual.

SECONDARY OUTCOMES:
PROMIS Short Form Depression | Past 7 days prior to completion of survey
  PROMIS Short Form Depression will measure distress on a 1 (never) to 5 (always) scale with lower scores denoting better outcome on a 5-point likert-type scale. Higher scores reflect higher distress.
Prognosis Treatment and Perceptions Questionnaire | Day 1 of completion of survey
  Prognosis Treatment and Perceptions Questionnaire will measure the treatment expectations and prognostic understanding using 8 items with varied response options..

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Steffen, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Laurie E Steffen, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Steffen McLouth LE, Lycan TW Jr, Levine BJ, Gabbard J, Ruiz J, Farris M, Grant SC, Pajewski NM, Weaver KE, Petty WJ. Patient-Reported Outcomes From Patients Receiving Immunotherapy or Chemoimmunotherapy for Metastatic Non-Small-Cell Lung Cancer in Clinical Practice. Clin Lung Cancer. 2020 May;21(3):255-263.e4. doi: 10.1016/j.cllc.2019.11.015. Epub 2019 Nov 29. PMID 31917067
- [Derived] McLouth LE, Gabbard J, Levine BJ, Golden SL, Lycan TW, Petty WJ, Weaver KE. Prognostic Awareness, Palliative Care Use, and Barriers to Palliative Care in Patients Undergoing Immunotherapy or Chemo-Immunotherapy for Metastatic Lung Cancer. J Palliat Med. 2023 Jun;26(6):831-836. doi: 10.1089/jpm.2022.0352. Epub 2023 Mar 13. PMID 36912809